CLINICAL TRIAL: NCT00189267
Title: Vehicle-Controlled, Double-Blind Study to Assess the Safety and Efficacy of Imiquimod 5% Cream Applied Once Daily 3 Days Per Week for the Treatment of Actinic Keratoses in Immunosuppressed Organ Transplant Recipients.
Brief Title: A Study to Evaluate the Effectiveness and Safety of Multiple Applications of Imiquimod 5% Cream for the Treatment of Actinic Keratoses in Organ Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1443-IMIQ
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2006-08

CONDITIONS: Actinic Keratosis
Keywords: Aldara; Actinic Keratosis; Graft Recipients
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

INTERVENTIONS:
Drug: Imiquimod 5 % Cream

SUMMARY:
The purpose of the study is to compare effectiveness and safety of multiple applications of imiquimod 5% cream and vehicle cream in graft recipients suffering from actinic keratosis.

ELIGIBILITY:
Inclusion Criteria:

* Have a total of 4-10 actinic keratosis (AK) lesions located on either face or scalp
* If female and of childbearing potential, have a negative urine pregnancy test at treatment initiation, and willing to use a medically acceptable method of contraception during the treatment period
* Renal, liver or heart transplant recipients

Exclusion Criteria:

* Graft rejection with loss of the graft in the medical history
* Unstable status of organ transplant disease during the last 12 months
* Known to be pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2002-11; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome of the study is to compare imiquimod 5% cream and vehicle cream with respect to safety assessments in graft recipients.

SECONDARY OUTCOMES:
Secondary outcome of the study is to compare imiquimod 5% cream and vehicle cream with respect to complete and partial clearance rates.

CONTACTS AND LOCATIONS:
Overall Officials: Study Coordinator, Study Chair — Universitaetsklinikum Charite